CLINICAL TRIAL: NCT04728282
Title: Randomized Clinical Trial Comparing Lateralized Reverse Total Shoulder Arthroplasty (RTSA) With and Without Subscapularis Repair
Brief Title: Comparison of Lateralized RTSA With and Without Subscapularis Repair
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Panam Clinic (Other)
Collaborators: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RSASUB-16-01-2021
Record Dates: First submitted 2021-01-22; First posted 2021-01-28 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Arthritis Shoulder
Keywords: reverse total shoulder arthroplasty; subscapularis; repair

STUDY DESIGN:
Intervention Model Description: This is a double-blinded randomized clinical trial comparing two groups, RTSA with and RTSA without subscapularis repair. Eighty-four participants will be randomized at a 1:1 ratio in blocks of 12. All participants will be recruited from the patient populations of six fellowship trained upper extremity orthopaedic surgeons at initial consult. Patients will be randomized intraoperatively using a telephone/web-based system.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients will be blinded to their group allocation. This is possible because the incision and rehabilitation processes are consistent between groups. It is not possible for the treating surgeon to be blinded to group allocation, therefore a research team member (athletic or physical therapist) will remain blinded to group allocation and conduct all study related assessments as well as administer the patient-reported questionnaires. This will be maintained by the participant not removing their shirt during the study assessment. Patients will not be informed of which procedure they will undergo until the study is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RTSA with subscapularis repair (Experimental)
  Interventions: Procedure: RTSA with subscapularis repair
- RTSA without subscapularis repair (Active Comparator)
  Interventions: Procedure: RTSA without subscapularis repair

INTERVENTIONS:
Procedure: RTSA with subscapularis repair — Lateralized reverse total shoulder arthroplasty with repair of subscapularis
  Arms: RTSA with subscapularis repair
Procedure: RTSA without subscapularis repair — Lateralized reverse total shoulder arthroplasty without repair of subscapularis
  Arms: RTSA without subscapularis repair

SUMMARY:
The purpose of this double-blind randomized controlled trial is to compare patient-reported, clinical, and functional outcomes in patients undergoing RTSA with and without subscapularis repair after placement of a modern "lateralized" implant over the course of 24-months postoperative.

DETAILED DESCRIPTION:
The main objective of this study is to compare patient-reported outcome measures (PROMs), and clinical and functional outcomes between RTSA with and without subscapularis repair. The specific aims for this study are:

Specific Aim 1:

To determine if there is a difference in PROM scores between RTSA with and without subscapularis repair during the 24-month postoperative period.

Specific Aim 2:

To determine if there is a difference between the two surgical approaches with respect to shoulder function, specifically range of motion and strength, during the 24-month postoperative period.

Specific Aim 3:

To determine if there is a difference in shoulder dislocation rates between RTSA with and without subscapularis repair during the 24-month postoperative period.

Specific Aim 4:

To determine if there is a difference in surgical complications, re-operation or revision rates between RTSA with and without subscapularis repair during the 24-month postoperative period.

Specific Aim 5:

To quantify the operative times for RTSA with and without subscapularis repair, and determine if there is a difference between the two approaches.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of glenohumeral arthritis, rotator cuff arthropathy, or massive irreparable rotator cuff tear with surgeon-patient decision to undergo RTSA
* First RTSA implantation
* Absence of neoplastic diseases at the treated site
* Fatty infiltration of the subscapularis is low-grade (i.e. Goutallier < Grade 3) based on pre-operative CT performed as standard of care in the patient group

Exclusion Criteria:

* Previous shoulder arthroplasty (hemi-, total shoulder, or RTSA)
* Avascular necrosis
* Post-infectious arthritis
* Proximal humerus fracture
* Inflammatory arthritis
* Inability to communicate in English
* Unable to return for study visits to 24-months post-operative (e.g. unable to arrange transportation to study appointments, plans to relocate, etc.)

Intra-operative Exclusions:

* Subscapularis with fatty infiltration (Goutallier ≥ 3)
* Subscapularis that is deemed to be irreparable. An irreparable tendon is defined as one that is not of sufficient quality or does not allow adequate excursion to reach the repair site
* Any anatomical or patient characteristic that warrants a non-lateralized implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
ASES Score | 24 months post-operative
  The ASES is a patient-reported upper extremity-specific functional assessment tool and is scored out of a maximum 100 points, where 100 represents maximum function and no pain (Richards et al., 1994). It has a pain component measured on a visual analog scale as well as ten Likert-scale questions on function (e.g., put on a coat, sleep on affected side). The ASES is reliable and is validated for this population and is one of the most commonly used shoulder outcomes in North America.

SECONDARY OUTCOMES:
Constant Score | baseline pre-operative
  The Constant Score is validated and reliable PROM/clinical tool used to evaluate overall shoulder function based on pain, activities of daily living, and the clinical evaluation of ROM and strength (Constant & Murley, 1987). This score is widely reported in European-based literature. Minimum value is 0 and maximum value is 100, with higher scores being a better outcome.
Constant Score | 3 months post-operative
  The Constant Score is validated and reliable PROM/clinical tool used to evaluate overall shoulder function based on pain, activities of daily living, and the clinical evaluation of ROM and strength (Constant & Murley, 1987). This score is widely reported in European-based literature. Minimum value is 0 and maximum value is 100, with higher scores being a better outcome.
Constant Score | 6 months post-operative
  The Constant Score is validated and reliable PROM/clinical tool used to evaluate overall shoulder function based on pain, activities of daily living, and the clinical evaluation of ROM and strength (Constant & Murley, 1987). This score is widely reported in European-based literature. Minimum value is 0 and maximum value is 100, with higher scores being a better outcome.
Constant Score | 12 months post-operative
  The Constant Score is validated and reliable PROM/clinical tool used to evaluate overall shoulder function based on pain, activities of daily living, and the clinical evaluation of ROM and strength (Constant & Murley, 1987). This score is widely reported in European-based literature. Minimum value is 0 and maximum value is 100, with higher scores being a better outcome.
Constant Score | 24 months post-operative
  The Constant Score is validated and reliable PROM/clinical tool used to evaluate overall shoulder function based on pain, activities of daily living, and the clinical evaluation of ROM and strength (Constant & Murley, 1987). This score is widely reported in European-based literature. Minimum value is 0 and maximum value is 100, with higher scores being a better outcome.
SANE Score | baseline pre-operative
  The Single Assessment Numeric Evaluation (SANE) score is a single question that asks patients to rate their affected shoulder as a percentage of normal to provide a simple and efficient measure of patient outcome (Gowd et al., 2019). Patients will be asked the following question: "How would you rate your affected shoulder today as a percentage of normal (0% to 100% scale with 100% being normal)?"
SANE Score | 3 months post-operative
  The Single Assessment Numeric Evaluation (SANE) score is a single question that asks patients to rate their affected shoulder as a percentage of normal to provide a simple and efficient measure of patient outcome (Gowd et al., 2019). Patients will be asked the following question: "How would you rate your affected shoulder today as a percentage of normal (0% to 100% scale with 100% being normal)?"
SANE Score | 6 months post-operative
  The Single Assessment Numeric Evaluation (SANE) score is a single question that asks patients to rate their affected shoulder as a percentage of normal to provide a simple and efficient measure of patient outcome (Gowd et al., 2019). Patients will be asked the following question: "How would you rate your affected shoulder today as a percentage of normal (0% to 100% scale with 100% being normal)?"
SANE Score | 12 months post-operative
  The Single Assessment Numeric Evaluation (SANE) score is a single question that asks patients to rate their affected shoulder as a percentage of normal to provide a simple and efficient measure of patient outcome (Gowd et al., 2019). Patients will be asked the following question: "How would you rate your affected shoulder today as a percentage of normal (0% to 100% scale with 100% being normal)?"
SANE Score | 24 months post-operative
  The Single Assessment Numeric Evaluation (SANE) score is a single question that asks patients to rate their affected shoulder as a percentage of normal to provide a simple and efficient measure of patient outcome (Gowd et al., 2019). Patients will be asked the following question: "How would you rate your affected shoulder today as a percentage of normal (0% to 100% scale with 100% being normal)?"
EQ5D-3L | baseline, pre-operative
  The EQ-5D is valid, reliable, responsive PROM used to document overall wellness based on 5 dimensions: mobility, self-care, usual activities, pain, anxiety/depression (Herdman et al., 2011). A single value is calculated (the value index), which indicates how good or bad a patient's health state is relative to a specified population. There are two components, VAS for general health, with 0 minimum and 100 maximum, with higher scores being more positive. The second component is a 25 point scale with minimum 5 and maximum 25 wit h lower scores more positive.
EQ5D-3L | 3 months, post-operative
  The EQ-5D is valid, reliable, responsive PROM used to document overall wellness based on 5 dimensions: mobility, self-care, usual activities, pain, anxiety/depression (Herdman et al., 2011). A single value is calculated (the value index), which indicates how good or bad a patient's health state is relative to a specified population. There are two components, VAS for general health, with 0 minimum and 100 maximum, with higher scores being more positive. The second component is a 25 point scale with minimum 5 and maximum 25 wit h lower scores more positive.
EQ5D-3L | 6 months, post-operative
  The EQ-5D is valid, reliable, responsive PROM used to document overall wellness based on 5 dimensions: mobility, self-care, usual activities, pain, anxiety/depression (Herdman et al., 2011). A single value is calculated (the value index), which indicates how good or bad a patient's health state is relative to a specified population. There are two components, VAS for general health, with 0 minimum and 100 maximum, with higher scores being more positive. The second component is a 25 point scale with minimum 5 and maximum 25 wit h lower scores more positive.
EQ5D-3L | 12 months, post-operative
  The EQ-5D is valid, reliable, responsive PROM used to document overall wellness based on 5 dimensions: mobility, self-care, usual activities, pain, anxiety/depression (Herdman et al., 2011). A single value is calculated (the value index), which indicates how good or bad a patient's health state is relative to a specified population. There are two components, VAS for general health, with 0 minimum and 100 maximum, with higher scores being more positive. The second component is a 25 point scale with minimum 5 and maximum 25 wit h lower scores more positive.
EQ5D-3L | 24 months, post-operative
  The EQ-5D is valid, reliable, responsive PROM used to document overall wellness based on 5 dimensions: mobility, self-care, usual activities, pain, anxiety/depression (Herdman et al., 2011). A single value is calculated (the value index), which indicates how good or bad a patient's health state is relative to a specified population. There are two components, VAS for general health, with 0 minimum and 100 maximum, with higher scores being more positive. The second component is a 25 point scale with minimum 5 and maximum 25 wit h lower scores more positive.
Range of Motion | baseline, pre-surgery
  For both shoulders, forward flexion and external rotation at 0 and 90 degrees abduction will be measured with a goniometer and reported in degrees.
Range of Motion | 3 months, post-operative
  For both shoulders, forward flexion and external rotation at 0 and 90 degrees abduction will be measured with a goniometer and reported in degrees.
Range of Motion | 6 months, post-operative
  For both shoulders, forward flexion and external rotation at 0 and 90 degrees abduction will be measured with a goniometer and reported in degrees.
Range of Motion | 12 months, post-operative
  For both shoulders, forward flexion and external rotation at 0 and 90 degrees abduction will be measured with a goniometer and reported in degrees.
Range of Motion | 24 months, post-operative
  For both shoulders, forward flexion and external rotation at 0 and 90 degrees abduction will be measured with a goniometer and reported in degrees.
Isometric Strength | baseline, pre-surgery
  Measured using a hand-held dynamometer, in flexion, abduction, and external rotation
Isometric Strength | 3 months, post-operative
  Measured using a hand-held dynamometer, in flexion, abduction, and external rotation
Isometric Strength | 6 months, post-operative
  Measured using a hand-held dynamometer, in flexion, abduction, and external rotation
Isometric Strength | 12 months, post-operative
  Measured using a hand-held dynamometer, in flexion, abduction, and external rotation
Isometric Strength | 24 months, post-operative
  Measured using a hand-held dynamometer, in flexion, abduction, and external rotation
ASES Score | baseline, pre-operative
  The ASES is a patient-reported upper extremity-specific functional assessment tool and is scored out of a maximum 100 points, where 100 represents maximum function and no pain (Richards et al., 1994). It has a pain component measured on a visual analog scale as well as ten Likert-scale questions on function (e.g., put on a coat, sleep on affected side). The ASES is reliable and is validated for this population and is one of the most commonly used shoulder outcomes in North America.
ASES Score | 3 months, post-operative
  The ASES is a patient-reported upper extremity-specific functional assessment tool and is scored out of a maximum 100 points, where 100 represents maximum function and no pain (Richards et al., 1994). It has a pain component measured on a visual analog scale as well as ten Likert-scale questions on function (e.g., put on a coat, sleep on affected side). The ASES is reliable and is validated for this population and is one of the most commonly used shoulder outcomes in North America.
ASES Score | 6 months, post-operative
  The ASES is a patient-reported upper extremity-specific functional assessment tool and is scored out of a maximum 100 points, where 100 represents maximum function and no pain (Richards et al., 1994). It has a pain component measured on a visual analog scale as well as ten Likert-scale questions on function (e.g., put on a coat, sleep on affected side). The ASES is reliable and is validated for this population and is one of the most commonly used shoulder outcomes in North America.
ASES Score | 12 months, post-operative
  The ASES is a patient-reported upper extremity-specific functional assessment tool and is scored out of a maximum 100 points, where 100 represents maximum function and no pain (Richards et al., 1994). It has a pain component measured on a visual analog scale as well as ten Likert-scale questions on function (e.g., put on a coat, sleep on affected side). The ASES is reliable and is validated for this population and is one of the most commonly used shoulder outcomes in North America.

CONTACTS AND LOCATIONS:
Overall Officials: Jarret Woodmass, MD, Principal Investigator — Pan Am Clinic
Locations (1):
- Pan Am Clinic, Winnipeg, Manitoba, Canada